CLINICAL TRIAL: NCT06623747
Title: Low Energy Availability and Recovery From Resistance Exercise
Acronym: LEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chaise Murphy (Other)
Collaborators: South Dakota State University (Other)
Responsible Party: Sponsor-Investigator, Chaise Murphy, Assistant Professor of Exercise Science, South Dakota State University
Organization: South Dakota State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB-2024-43
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Resistance Exercise
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL (Active Comparator)
  Interventions: Behavioral: Diet
- LOW ENERGY AVAILABILITY (Experimental)
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — 15 kcal per kg fat-free mass
  Arms: LOW ENERGY AVAILABILITY
Behavioral: Diet — 45 kcal per kg fat-free mass
  Arms: CONTROL

SUMMARY:
This research project will determine how restricting Calories to lose weight affects your ability to recover between weightlifting exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

* 3 years of resistance training experience

Exclusion Criteria:

* 1+ American College of Sports Medicine sign(s) or symptom(s) of cardiovascular, metabolic or renal disease(s)
* musculoskeletal disorder(s)
* lactose intolerance; soy or dairy allergies

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Performance | At enrollment (baseline), wait 1-2 weeks, before and after first 2-day condition, wait 1-2 weeks, before and after second 2-day condition
Knee Extension and Flexion Repetitions to Failure | At enrollment (baseline), wait 1-2 weeks, before and after first 2-day condition, wait 1-2 weeks, before and after second 2-day condition
Bench Press One-Repetition Maximum | At enrollment (baseline), wait 1-2 weeks, before and after first 2-day condition, wait 1-2 weeks, before and after second 2-day condition
Peak Knee Extension and Flexion Torques | At enrollment (baseline), wait 1-2 weeks, before and after first 2-day condition, wait 1-2 weeks, before and after second 2-day condition

CONTACTS AND LOCATIONS:
Overall Officials: Chaise A Murphy, Ph.D., Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Brookings, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
As of right now, I have no collaborators to share the data with.